CLINICAL TRIAL: NCT03752099
Title: A Phase 1b/2 Study to Evaluate the Safety and Tolerability of VERU-111 in Men With Advanced Metastatic Castration Resistant Prostate Cancer
Brief Title: To Evaluate Safety and Tolerability of VERU-111 in Men With Advanced Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: V1011101
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
MeSH Terms: interventions — sabizabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- VERU-111 4.5mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111
- VERU-111 9mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111
- VERU-111 18mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111
- VERU-111 27mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111
- VERU-111 36mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111
- VERU-111 45mg (Experimental): Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
  Interventions: Drug: VERU-111

INTERVENTIONS:
Drug: VERU-111 — VERU-111
  Other Names: Bisindole

SUMMARY:
Phase 1b - To assess the safety/tolerability of VERU-111 and to determine the maximum tolerated dose of VERU-111 in patients with metastatic, castration resistant prostate cancer who have failed a novel androgen blocking agent therapy (mCRPC).

Phase 2 - To estimate the PSA50 response rate, defined as a decline in PSA to ≥50% of baseline level, confirmed with a second measurement at least 3 weeks apart (PCWG3).

DETAILED DESCRIPTION:
Up to 7 sites in the US only with approximately 18 patients for Phase 1b portion (3 patients per dose group) of the study. Additional patients may be enrolled into the Phase 1b portion of the study depending on the safety and tolerability assessment in the dose escalation scheme.

Approximately 26 patients will be enrolled in the Phase 2 portion of the study

Phase 1b Approximately 18 patients for Phase 1b portion (3 patients per dose group) will be enrolled into the study. Additional subjects may be enrolled based on the assessment of safety and tolerability in the dose escalation scheme.

VERU-111 will be administered orally for three 21-day cycles in which the patient will take the study drug (capsules) daily with food for 7 days and then have a 14-day treatment free period.

Dose Escalation Criteria In Phase 1b, three patients will be planned at each dose level and followed for one 21-day cycle.

* If 0/3 patients exhibit a dose limiting toxicity (DLT) after one 21-day cycle, the next patient will be treated at the next dose level.
* If one patient out of the 3 exhibits a DLT related to the study agent, the cohort will be expanded to up to 6 patients. If 1 of 6 patients exhibits a DLT related to the study agent, then the next patient will enroll at the next dose level.
* If 2 of the first 3 subjects OR 2 of the first 6 patients exhibit a DLT related to the study agent, the MTD is considered to have been determined and at least 3 additional patients will be entered at the dose level below the one at which DLT is observed. Dose escalations will occur no sooner than 3 weeks after the last patient on the dose level has begun therapy to allow for full assessment of DLT. No intra-patient escalation will be allowed.
* If <1 of 6 patients experience a DLT, this will be the recommended Phase 2 dose for the expansion cohorts.

A Cohort Review Committee, consisting of investigators, the medical monitor and the sponsor, will monitor the trial on an ongoing basis for safety and will guide dose escalation decisions based on the occurrence of DLTs as described in this protocol.

The planned dosing for VERU-111 in the Phase 1b portion will be:

Treatment Group Daily dose Dosing Regimen

1. 4.5mg Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
2. 9mg Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
3. 18mg Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
4. 27mg Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
5. 36mg Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.
6. 45mg1 Daily dosing on Day 1-7 of each 21-day cycle for 3 cycles Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.Treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.

1 If after the first 21-day cycle for the 45 mg in Treatment Group 5 no DLT is observed, then additional dose levels and additional dosing schedules (i.e. 14 days of daily dosing followed by a 7-day treatment free period) may be considered.

Phase 2 The maximum tolerated dose of VERU-111 identified in the Phase 1b portion of the study will be used in the Phase 2 portion of the study. The dosing regimen will be daily dosing for 7 days followed by a 14-day treatment free period (21-day cycle). Three 21-day cycles are planned in this study. However, treatment may continue past the planned three 21-day cycles until DLT or disease progression is observed.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, patients should meet all of the following criteria:

• Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Patients >18 years of age.
* Histological or cytologic proof of adenocarcinoma of the prostate.
* Radiographic evidence of metastatic disease by CT scan or MRI and/or bone scan.
* Known castration resistant prostate cancer, defined according to PCWG3 criteria.
* Subjects who have metastatic castration resistant prostate cancer that have maintained ADT and have failed a novel androgen receptor agent (abiraterone or enzalutamide) defined as:

  * Serum PSA progression of two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least two weeks apart.

Or

* Documented bone lesions by the appearance of two or more new lesions on bone scintigraphy or dimensionally-measurable soft tissue metastatic lesion assessed by CT or MRI.

  * Absolute PSA ≥2.0 ng/ml at screening.
  * Prior chemotherapy for mCRPC:
* Phase 1b - ONE prior taxane chemotherapy for mCRPC will be allowed during the Phase 1b portion of study as long as the last dose was more than four weeks prior to the first dose of study drug.
* Phase 2 - Prior chemotherapy for mCRPC is not allowed in the Phase 2 portion of the study. Prior chemotherapy for metastatic hormone sensitive prostate cancer will not qualify as a prior chemotherapy and the last dose must be >6 months prior to enrollment.

  * Prior treatment with abiraterone, enzalutamide, bicalutamide, and/or ketoconazole is allowed. There is no limit on the maximum number or types of prior hormonal therapies received. The patients should be off prior therapy for at least two weeks (4 weeks off bicalutamide or nilutamide treatment) prior to first dose of study drug.
  * ECOG performance status ≤2.
  * Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Hemoglobin 9.0 g/dL with no blood transfusion in the past 28 days.
* Absolute neutrophil count (ANC) 1.5 x 109/L.
* Platelet count 100 x 109/L.
* Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) (or <2.5 x ULN for patients with known Gilberts disease).
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT))/Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤2.5 x institutional upper limit of normal.

Note: Patients with elevations in bilirubin, AST, or ALT should be thoroughly evaluated for the etiology of this abnormality prior to entry and patients with evidence of viral infection should be excluded.

* Participants must have a life expectancy >3 months.
* Male participants, and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination [see Appendix E for acceptable methods], throughout the period of taking study treatment and for at least 4 weeks after the last dose of VERU-111 to prevent pregnancy in a partner.
* Other than the metastatic prostate cancer, no evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin or other cancers treated with curative intent >3 years prior).
* Participants must agree to either refrain from prolonged exposure to the sun or agree to use at least SPF 50 on all exposed skin and protective clothing during prolonged sun exposure throughout participation in this study and/or treatment with VERU-111.

Exclusion Criteria:

Patients that meet any of the criteria listed below will not be eligible for study entry:

* Histologic identification of small cell carcinoma of the prostate or neuroendocrine pathology in either biopsy or prostatectomy tissue.
* Has received external-beam radiotherapy within the last 2 weeks prior to start of study treatment.
* Patients receiving full dose anticoagulation therapy are not eligible for study.
* Patients with prior history of a thromboembolic event within the last 6 months.
* Participation in another clinical study with an investigational product during the last 4 weeks/28 days.
* Patients should be excluded if they have had prior systemic treatment with two prior taxane chemotherapies for advanced prostate cancer. No limit to other prior therapies.
* Concurrent use of other anticancer agents (see Appendix G) or treatments, with the following exceptions:

  o Ongoing treatment with denosumab (Prolia) or bisphosphonate (e.g., zoledronic acid) is allowed. Ongoing treatment should be kept at a stable schedule; however, if medically required, a change of dose, compound, or both is allowed.
* Any treatment modalities involving major surgery within 4 weeks prior to the start of study treatment.
* Patients are excluded if they have active known brain metastases or leptomeningeal metastases.
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* History of severe hypersensitivity reaction to any taxane chemotherapy.
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.
* Total bilirubin levels > ULN or OR AST/ALT levels >1.5xULN with WITH concomitant alkaline phosphatase levels >2.5xULN.

The following exclusion criterion is added to the Phase 1b portion of the study only:

• Patients with substantial visceral disease who require immediate treatment with cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 21 Days
  Patients will be assessed for toxicities at each clinical evaluation. Toxicities will be graded according to CTCAE v5.0 standardized grading scales. The incidence of grade 3-5 toxicities will be reported.Toxicities will be reported as a tabulated table by type and grade.
PSA50 Response Rate | 63 Days
  Decrease in the PSA to ≥50% less than the baseline PSA upon enrollment in the trial. The decrease must be confirmed by a second measurement at least 3 weeks apart. PSA values will be measured monthly during the trial. All patients who take at least one dose of VERU-111 will be considered evaluable for the primary endpoint. If patients do not have at least one follow-up PSA after initiation of VERU-111 due to stopping therapy for toxicity or withdrawing consent, then they will be replaced. PSA50 response rate will be estimated along with 95% confidence interval.

SECONDARY OUTCOMES:
PSA progression-free survival | 63 Days
  PSA progression per PCWG3 will be used. PSA-PFS will be defined as an increase in 25% over a nadir value, confirmed by a follow-up PSA at least 3 weeks later. If patients are removed from study prior to PSA progression, then they will be censored at that time. We will use the Kaplan-Meier method to summarize the median PSA-PFS.
Progression-free survival | 63 days
  Measured from the time of first dose to objective clinical or radiographic tumor progression as defined by PCWG3 for progressive disease or death and summarized using a Kaplan-Meier curve. The time to progression will be the earliest observed time of progression. Patients whose disease has not progressed at follow-up will either be censored at the date of follow-up or if they continue therapy after the planned 3 cycles, they will be followed for progression. A Kaplan-Meier method will be used to summarize the median PFS.
Percentage of Patients who achieve Objective Response Rate | 63 Days
  Percentage of patients who achieve an objective response by RECIST1.1 criteria (i.e. Complete response or Partial Response) to VERU-111. The objective response rate and the exact 95% confidence interval will be estimated for the population of patients with RECIST evaluable disease.
Number of participants with treatment related adverse events (Safety and Tolerability) | 91 Days
  Standard safety summaries will be provided for treatment exposure, patient disposition, adverse events leading to discontinuation, serious adverse events, and all events resulting in death, including those up to 28 days after treatment discontinuation. The incidence of adverse events will be tabulated and reviewed for potential significance and clinical importance using CTCAE v5.0 grade ≥3 toxicities experienced by patients on the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.
Locations (13):
- United States (13):
  - Colorado Urology, Golden, Colorado
  - Universal Axon, Miami, Florida
  - First Urology, Jeffersonville, Indiana
  - Regional Urology, Shreveport, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Chesapeake Urology, Towson, Maryland
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Sargon Research, Canton, Ohio
  - Urologic Consultants, Bala-Cynwyd, Pennsylvania
  - Urology Clinics of North Texas, Dallas, Texas
  - Research Network America, Houston, Texas
  - Urology San Antonio, San Antonio, Texas
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Undecided